CLINICAL TRIAL: NCT04177511
Title: Treatment of Chronic Pelvic Pain Due to Endometriosis by Transcutaneous Auricular Vagus Nerve Stimulation
Acronym: Stim-Endom
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Hopital Foch (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2019-0057
Record Dates: First submitted 2019-11-13; First posted 2019-11-26 (Actual); Last update posted 2025-11-21 (Actual); Status verified 2025-11

CONDITIONS: Endometriosis
Keywords: Chronic pelvic pain; Transcutaneous Auricular Vagus Nerve Stimulation
MeSH Terms: conditions — Endometriosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Transcutaneous auricular vagus nerve stimulation (Experimental): A 30-minute session twice a day during 3 months of transcutaneous auricular vagus nerve stimulation using the TENS Eco Plus.
  Standard treatment will be continued by the patients of this arm.
  Interventions: Device: Transcutaneous Auricular Vagus Nerve Stimulation
- Standard treatment (No Intervention): Patients of this arm will continue their standard treatment.

INTERVENTIONS:
Device: Transcutaneous Auricular Vagus Nerve Stimulation — Transcutaneous Auricular Vagus Nerve Stimulation has an eartip connected to an external stimulator. The device used in this study is the TENS Eco Plus commercialized by Schwa Medico and European Compliance (CE) marked.
  The electrode is positioned in the cymba concha of the left ear.
  Arms: Transcutaneous auricular vagus nerve stimulation

SUMMARY:
6-10% of women of childbearing age suffer from endometriosis, which is mainly manifested by dysmenorrhea, non-menstrual pelvic pain and dyspareunia. Several treatment strategies, including surgical ones, are proposed but they are sometimes insufficient because endometriosis-related pain is frequently accompanied by sensitization. Endometriosis surgery, when indicated, is therefore changeably effective, even though the lesions have been completely resected. Patients therefore consult Pain Units seeking for the effective treatment as the pain persist even after surgical management of endometriosis.

Vagus nerve stimulation is a non-invasive technique that includes an anti-inflammatory effect and a modulation of neurotransmitter production (adrenaline, norepinephrine; serotonin, acetylcholine). Yuan and Silberstein published a general review on the technique. Migraine and depression are one of the selected indications. In addition, Napadow et al. published favourable results in a short series of patients with chronic pelvic pain. The Investigators of this study have treated some patients with this technique with a result deemed satisfactory which leads to propose a randomized study to confirm this impression.

ELIGIBILITY:
Inclusion Criteria:

* Women aged >= 15 years
* With chronic pelvic pain and/ or dysmenorrhoea and/ or dyspareunia
* Who has been cared for by a gynecologist in one of the institutions participating in the study
* Diagnosed with endometriosis
* Having signed an informed written consent
* Affiliated to a health insurance scheme

Exclusion Criteria:

* contraindication to the use of transcutaneous auricular vagus nerve stimulation (cardiac pathology, asthmatic patient)
* pregnant or breastfeeding women
* patient undergoing in vitro fertilization
* associated pathology requiring long-term analgesic treatment
* patient with atria trans vagal neurostimulation in the 12 months prior to inclusion
* patient deprived of liberty or under guardianship

Min Age: 15 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 72 (Estimated)
Dates: Start 2021-12-13 (Actual); Primary Completion 2027-03-28 (Estimated); Study Completion 2027-03-28 (Estimated)

PRIMARY OUTCOMES:
Change of symptoms related to the pelvic pain | 3 months after enrolment
  Self assessement of change using Patient's Global Impression of Change (PGIC) scale in which patients rate the improvement of their symptoms related to their pelvic pain from "No change or it get worse" to "A great deal better, and a considerable improvement that has made all the difference" . A favorable result will be "Better, and a definite improvement that has made a real and worthwhile difference" or "A great deal better, and a considerable improvement that has made all the difference"

SECONDARY OUTCOMES:
Efficacy on pain | Day 1 and 3 months after enrolment
  Self assessement of pain using Endometriosis-associated pelvic pain scale on which patients rate their current pain intensity from 0 "No pain" to 10 "worst possible pain"
Efficacy on severity of patient's symptoms | Day 1 and 3 months after enrolment
  Physician assessement of severity of patient's symptoms using Global Clinical Impressions-Severity scale on which physicians rate the severity of patient's symptoms from "not evaluated" to "Among the sickest patients"
Efficacy on quality of life | Day 1 and 3 months after enrolment
  Self assessement of quality of life using Endometriosis Health Profile-5
Efficacy on quality of life | Day 1 and 3 months after enrolment
  Self assessement of quality of life using EQ-5D scale
Efficacy on Anxiety | Day 1 and 3 months after enrolment
  Self assessement of anxiety using the Hospital Anxiety and Depression scale
Efficacy on gynecological and pelvic pain symptoms | Day 1 and 3 months after enrolment
  Self assessement of gynecological and pelvic pain symptoms using ENDOL-4D questionnaire
Efficacy on gynecological and pelvic pain symptoms | D1 and 3 months after enrolment
  Self assessement of gynecological and pelvic pain symptoms using KESS questionnaire
General efficacy of the device Transcutaneous Electronic Neuro Stimulation TENS Eco Plus | 3 months after enrolment
  Self assessement of satisfaction using a satisfaction questionnaire involving satisfaction, adherence to treatment sessions and ease of use of the device
Collection of possible side effects | 3 months after Enrolement
  collection of vagal malaise, nausea and vomiting

CONTACTS AND LOCATIONS:
Overall Officials: Mireille MICHEL-CHERQUI, MD, Principal Investigator — Hopital Foch, Suresnes; Marc FISCHLER, MD PhD, Study Chair — Hopital Foch, Suresnes
Locations (1):
- Hopital Foch, Suresnes, Île-de-France Region, France

IPD SHARING:
Plan to Share IPD: No